CLINICAL TRIAL: NCT01360853
Title: A Phase III, Multi-center, Randomized, Controlled Study to Compare the Efficacy and Safety of Gemcitabine Alone vs. ON 01910.Na Combined With Gemcitabine in Patients With Previously Untreated Metastatic Pancreatic Cancer
Brief Title: Gemcitabine and ON 01910.Na in Previously Untreated Metastatic Pancreatic Cancer
Acronym: ONTRAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Collaborators: Academic GI Cancer Consortium (AGICC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-22; 11PAN01 (Other: Academic Oncology GI Cancer Consortium)
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: pancreatic cancer; gemcitabine; ON 01910.Na; rigosertib sodium
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ON 01910; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Combination (Experimental): Arm A: Gemcitabine, 1000 mg/m2 weekly for 3 weeks of a 4 week cycle, + ON 01910.Na, 1800 mg/m2 via 2 hr CIV infusions administered twice weekly for 3 weeks of a 4 week cycle.
  Interventions: Drug: ON 01910.Na; Drug: Gemcitabine
- Arm B: Gemcitabine only (Active Comparator): Arm B: Gemcitabine only, 1000 mg/m2 weekly for 3 weeks of a 4 week cycle.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: ON 01910.Na — ON 01910.Na, 1800 mg/m2 via 2 hr CIV infusions administered twice weekly for 3 weeks of a 4 week cycle.
  Other Names: rigosertib sodium
  Arms: Arm A: Combination
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 weekly for 3 weeks of a 4 week cycle.
  Other Names: Gemzar; Gemcitabine HCl
  Arms: Arm A: Combination
Drug: Gemcitabine — Gemcitabine, 1000 mg/m2 weekly for 3 weeks of a 4 week cycle.
  Other Names: Gemzar; Gemcitabine HCl
  Arms: Arm B: Gemcitabine only

SUMMARY:
The question being asked in this study is: Will patients with advanced pancreatic cancer live significantly longer if they are treated with a combination of Gemcitabine and ON 01910.Na than if they are treated with Gemcitabine alone? There are two parts to this study. In the first part of the study, patients with metastatic pancreatic cancer who have received no prior chemotherapy for this disease will be assigned by chance either to the group that will be treated with both Gemcitabine and ON 01910.Na (about 100 patients will be in this group) or, to the group that will be treated with Gemcitabine only (about 50 patients will be in this group). How long patients survive in the 2 groups will be compared. If it looks like there is no difference between the groups, the study will stop. If it looks like patients in the group that were treated with both Gemcitabine and ON 01910.Na survive longer, the study will continue into a second part where more patients will be treated in order to confirm and better understand the findings of the first part of the study.

DETAILED DESCRIPTION:
This will be a Phase III study with sample size recalculation after 100 events have occurred. The study will be open-label, randomized, controlled, multi-center and will be conducted at approximately 200 to 300 study sites (60 to 80 study sites in the first portion of the trial).

In the first portion of the study, a total of 150 patients with metastatic pancreatic cancer who have received no prior chemotherapy for this disease will be randomized in a 2:1 fashion to 1 of the 2 following treatment regimens:

* Arm A: Gemcitabine 1000 mg/m2 weekly for 3 weeks of a 4 week cycle + ON 01910.Na 1800 mg/m2 via 2 hr continuous intravenous infusion (CIV) infusions administered twice weekly for 3 weeks of a 4 week cycle (approximately 100 patients)
* Arm B: Gemcitabine only, 1000 mg/m2 weekly for 3 weeks of a 4 week cycle (approximately 50 patients).

Patients will be stratified at entry using the Eastern Cooperative Oncology Group (ECOG) performance status (ECOG scores of 0 1 vs. ECOG scores of 2; patients with higher scores will not be enrolled).

Patients will remain on study until disease progression or death from any cause, whichever comes first. Moreover, after treatment discontinuation for any cause, all patients will be followed until death.

After 150 patients have been enrolled, accrual will pause and patients will be followed until 100 deaths have occurred. At that time, the Data Safety Monitoring Committee (DSMC) will oversee a formal interim analysis to compare overall survival (OS) between the 2 groups and may recommend early stopping for futility. If the study continues after interim analysis, then the randomization scheme will continue up to 364 patients or the newly-calculated sample size. The maximum number of enrolled patients will be 650. The number of clinical sites may be expanded up to approximately 200 to 300 centers.

Patients in the gemcitabine-only arm (Arm B) will not be allowed to cross over to the combined treatment arm (Arm A). In addition, no palliative radiotherapy will be allowed during the trial.

The primary analysis will compare OS in the ON 01910.Na + gemcitabine arm (Arm A) vs. gemcitabine-only arm (Arm B) once an appropriate number of events has been reached. There are 2 secondary efficacy outcomes: progression-free survival (PFS) and objective response.

Toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v4.03. Grade 3 and 4 hematologic toxicities and > Grade 2 non-hematologic toxicities will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old presenting with histopathologically or cytologically confirmed metastatic adenocarcinoma of the pancreas; metastatic disease is defined as disease which has spread beyond the peri-pancreatic lymph nodes.
* Patients must have received no prior chemotherapy for pancreatic cancer, including adjuvant chemotherapy.
* Measurable disease, defined as lesions that can be accurately measured in at least 1 dimension with longest diameter (LD) ≥20 mm using conventional techniques or ≥10 mm with spiral computed tomography (CT) scan; measurable lymph nodes must be ≥15 mm in the short axis.
* ECOG Performance Status of 0, 1, or 2.
* Patients must have adequate renal function and serum creatinine ≤2.0 mg/dL.
* Patients must have adequate liver function as defined by total bilirubin ≤2.0 mg/dL and transaminase levels no higher than 3.0 times the institution's upper limit of normal (ULN). Patients with hepatic metastases may have transaminase levels of up to 5.0 times the ULN.
* All patients must have a serum albumin ≥3.0 g/dL.
* Patients must have adequate bone marrow (BM) function as defined by a granulocyte count ≥1,500/mm3, a platelet count ≥100,000/mm3, and hemoglobin >9 g/dL.
* Disease-free period of more than 5 years from prior malignancies other than pancreas (except curatively treated basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix and ductal carcinoma in situ [DCIS] breast disease).
* Adequate contraceptive regimen (including prescription oral contraceptives [birth control pills], contraceptive injections, intrauterine device [IUD], double-barrier method [spermicidal jelly or foam with condoms or diaphragm], contraceptive patch, or surgical sterilization) before entry and throughout the study for female patients of reproductive potential or female partners of male patients.
* Female patient with reproductive potential must have a negative urine beta human chorionic gonadotropin (bHCG) pregnancy test at Screening.
* Willing to adhere to the prohibitions and restrictions specified in this protocol.
* Patient must have signed an informed consent document.

Exclusion Criteria:

* Patients with unresectable locally advanced disease without evidence of disease elsewhere.
* Life expectancy of less than 12 weeks.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension or seizure disorder.
* Active infection not adequately responding to appropriate therapy.
* Symptomatic or clinically evident ascites.
* Serum sodium less than 130 mEq/L or conditions that may predispose patients to hyponatremia.
* Female patients who are pregnant or lactating.
* Male patients with female sexual partners who are unwilling to follow the strict contraception requirements described in this protocol.
* Major surgery without full recovery or major surgery within 3 weeks of ON 01910.Na treatment start.
* Evidence of brain metastases.
* Any concurrent administration and/or prior administration within 4 weeks of the first dose of study drug, of radiotherapy, or immunotherapy.
* Psychiatric illness/social situations that would limit the patient's ability to tolerate and/or comply with study requirements, or inability to comply with study and/or follow-up procedures (e.g., drug addition, chronic non-compliance, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-05; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Survival | 18 months
  This study's primary outcome is overall survival, defined as the time from randomization to death from any cause. All patients will be followed until death. Patients lost to follow-up will be censored at the time last known alive.

SECONDARY OUTCOMES:
Progression-free survival | 18 months
  Progression-free survival is defined as the time from the randomization to documented disease progression or death. Patients who are alive and do not have disease progression by the clinical cutoff will be censored at the dates of their last tumor evaluation. Kaplan-Meier curves for PFS will be compared using a stratified log-rank test (stratified by ECOG status: 0-1 vs. 2). Hazard ratios and 95% confidence intervals will be estimated using stratified Cox proportional hazards models.
Tumor size | 18 months
  Objective tumor response rates using Response Evaluation Criteria In Solid Tumors (RECIST).
Safety/tolerability | 18 months
  Toxicity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.03
QOL questionnaire | 18 months
  Quality of life (QOL) questionnaire, using the European Organisation for Research and Treatment of Cancer(EORTC) QLQ-C30 version 3.
Biomarkers | 18 months
  In this study, archival tissue will be collected and analyzed in order to identify molecular characteristics of pancreas tumors, which may confer susceptibility or resistance to gemcitabine alone or in combination with ON 01910.Na.
Population Pharmacokinetics | 18 months
  Measurement of ON 01910.Na in plasma of all patients in Arm A 1 hour after starting ON 01910.Na infusion at Day 1 and Day 15 in Cycle 1 only.
Full Pharmacokinetics | 18 Months
  At a limited number of sites, blood samples for measurement of ON 01910.Na and gemcitabine will be obtained at Cycle 1 Day 1 only, in a subset of 10 patients in Arm A, at the following 12 time-points: predose; 15 min after starting gemcitabine infusion; 30 min, immediately before ending gemcitabine infusion; 15 min after starting ON 01910.Na infusion; 30 min after ON 01910.Na infusion start; immediately before ending ON 01910.Na infusion; and, 15 min, 30 min, 1 hr, 2 hr, 4 hr and 8 hr after ending ON 01910.Na infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Wells Messersmith, MD, Study Chair — Anschutz Cancer Pavilion; Lawrence P. Leichman, MD, Study Chair — Academic Oncology Gastrointestinal Cancer Consortium; Antonio Jimeno, MD, PhD, Study Chair — Anschutz Cancer Pavilion
Locations (46):
- United States (30):
  - UCSD Moores Cancer Center, La Jolla, California
  - Desert Comprehensive Cancer Center, Palm Springs, California
  - Pacific Cancer Care, Salinas, California
  - Premiere Oncology, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Kaiser Permanente Colorado, Denver, Colorado
  - Poudre Valley Cancer Center of the Rockies, Fort Collins, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - University of Kansas Cancer Center, Westwood, Kansas
  - UMASS Medical School, Worcester, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Billings Clinic Cancer Center, Billings, Montana
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York University Langone Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Rex Cancer Center UNC Healthcare, Raleigh, North Carolina
  - St. Alexis Medical Center-Mid Dakota Clinic PC, Bismarck, North Dakota
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - Kaiser Permanente NW, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina - Hollings Cancer Center, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
- Hungary (3):
  - Semmelweis University Department of Diagnostic Radiology and Oncotherapy, Budapest
  - Semmelweis University, 3rd Department of Internal Medicine, Budapest
  - Hetenyi Geza Hospital 5004, Szolnok, Hungary, Szolnok
- India (6):
  - Basavatarakam Indo-American Cancer Hospital, Hyderabad, Andhra Pradesh
  - Regional Cancer Center, Thiruvananthapuram, Kerala
  - Jaslok Hospital & Research Centre, Mumbai, Maharashtra
  - Shatabdi Superspeciality Hospital, Nashik, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Lifeline Multispeciality Hospitals, Chennai, Tamil Nadu
- Russia (6):
  - State Budget Medical Institution of the Arkhangelsk Region, Arkhangelsk
  - Chelyabinsk Regional Clinical Oncology Center, Chelyabinsk
  - State Budget Medical Institution Clinical Oncology Center 1, Krasnodar
  - Budget Medical Institution of the Omsk Region: Clinical Oncology Center, Omsk
  - State Budget Medical Institution: Leningrad Regional Clinical Hospital, Saint Petersburg
  - State Medical Institution: Tula Regional Oncology Center, Tula
- Zakarpattia Regional Clinical Oncology Center Department of Chemotherapy, Uzhhorod, Ukraine

REFERENCES:
- [Background] Jimeno A, Chan A, Cusatis G, Zhang X, Wheelhouse J, Solomon A, Chan F, Zhao M, Cosenza SC, Ramana Reddy MV, Rudek MA, Kulesza P, Donehower RC, Reddy EP, Hidalgo M. Evaluation of the novel mitotic modulator ON 01910.Na in pancreatic cancer and preclinical development of an ex vivo predictive assay. Oncogene. 2009 Jan 29;28(4):610-8. doi: 10.1038/onc.2008.424. Epub 2008 Nov 24. PMID 19029951
- [Background] Jimeno A, Li J, Messersmith WA, Laheru D, Rudek MA, Maniar M, Hidalgo M, Baker SD, Donehower RC. Phase I study of ON 01910.Na, a novel modulator of the Polo-like kinase 1 pathway, in adult patients with solid tumors. J Clin Oncol. 2008 Dec 1;26(34):5504-10. doi: 10.1200/JCO.2008.17.9788. Epub 2008 Oct 27. PMID 18955447
- [Result] O'Neil BH, Scott AJ, Ma WW, Cohen SJ, Aisner DL, Menter AR, Tejani MA, Cho JK, Granfortuna J, Coveler AL, Olowokure OO, Baranda JC, Cusnir M, Phillip P, Boles J, Nazemzadeh R, Rarick M, Cohen DJ, Radford J, Fehrenbacher L, Bajaj R, Bathini V, Fanta P, Berlin J, McRee AJ, Maguire R, Wilhelm F, Maniar M, Jimeno A, Gomes CL, Messersmith WA. A phase II/III randomized study to compare the efficacy and safety of rigosertib plus gemcitabine versus gemcitabine alone in patients with previously untreated metastatic pancreatic cancer. Ann Oncol. 2016 Jun;27(6):1180. doi: 10.1093/annonc/mdw095. Epub 2016 Mar 3. No abstract available. PMID 26945010
- [Result] O'Neil BH, Scott AJ, Ma WW, Cohen SJ, Leichman L, Aisner DL, Menter AR, Tejani MA, Cho JK, Granfortuna J, Coveler L, Olowokure OO, Baranda JC, Cusnir M, Phillip P, Boles J, Nazemzadeh R, Rarick M, Cohen DJ, Radford J, Fehrenbacher L, Bajaj R, Bathini V, Fanta P, Berlin J, McRee AJ, Maguire R, Wilhelm F, Maniar M, Jimeno A, Gomes CL, Messersmith WA. A phase II/III randomized study to compare the efficacy and safety of rigosertib plus gemcitabine versus gemcitabine alone in patients with previously untreated metastatic pancreatic cancer. Ann Oncol. 2015 Dec;26(12):2505. doi: 10.1093/annonc/mdv477. Epub 2015 Oct 21. No abstract available. PMID 26489442
- [Result] O'Neil BH, Scott AJ, Ma WW, Cohen SJ, Aisner DL, Menter AR, Tejani MA, Cho JK, Granfortuna J, Coveler L, Olowokure OO, Baranda JC, Cusnir M, Phillip P, Boles J, Nazemzadeh R, Rarick M, Cohen DJ, Radford J, Fehrenbacher L, Bajaj R, Bathini V, Fanta P, Berlin J, McRee AJ, Maguire R, Wilhelm F, Maniar M, Jimeno A, Gomes CL, Messersmith WA. A phase II/III randomized study to compare the efficacy and safety of rigosertib plus gemcitabine versus gemcitabine alone in patients with previously untreated metastatic pancreatic cancer. Ann Oncol. 2015 Sep;26(9):1923-1929. doi: 10.1093/annonc/mdv264. Epub 2015 Jun 19. PMID 26091808
- See also: Related information about Academic Oncology Gastrointestinal Cancer Consortium (AGICC). — http://www.agicc.org